CLINICAL TRIAL: NCT01362764
Title: A Single-Dose, Open-Label, Randomized, Crossover Study to Assess the Relative Bioavailability of Two Abiraterone Acetate Suspension Formulations Compared to the Abiraterone Acetate Tablet Formulation Under Fasted Condition in Healthy Adult Subjects
Brief Title: A Study to Assess the Relative Bioavailability of Two Abiraterone Acetate Suspension Formulations Compared to the Abiraterone Acetate Tablet Formulation in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cougar Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CR018067; 212082HPL1001
Record Dates: First submitted 2011-05-27; First posted 2011-05-30 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Volunteers
Keywords: Abiraterone Acetate; ZYTIGA
MeSH Terms: interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Other): Abiraterone acetate tablets Type=exact unit=mg number= 250 form=tablet route=oral use as a single dose
  Interventions: Drug: Abiraterone acetate tablets
- 002 (Other): Abiraterone acetate suspension Formulation 1 Type=exact unit=mg/mL number=25 form=oral suspension route=oral use as a single dose of 10 mL
  Interventions: Drug: Abiraterone acetate suspension Formulation 1
- 003 (Other): Abiraterone acetate suspension Formulation 2 Type=exact unit=mg/mL number=25 form=oral suspension route=oral use as a single dose of 10 mL
  Interventions: Drug: Abiraterone acetate suspension Formulation 2

INTERVENTIONS:
Drug: Abiraterone acetate suspension Formulation 1 — Type=exact, unit=mg/mL, number=25, form=oral suspension, route=oral use, as a single dose of 10 mL
  Arms: 002
Drug: Abiraterone acetate suspension Formulation 2 — Type=exact, unit=mg/mL, number=25, form=oral suspension, route=oral use, as a single dose of 10 mL
  Arms: 003
Drug: Abiraterone acetate tablets — Type=exact, unit=mg, number= 250, form=tablet, route=oral use, as a single dose
  Arms: 001

SUMMARY:
The purpose of this study is to compare the single-dose pharmacokinetics (how the drug is absorbed in the body, distributed within the body, and how it is removed from the body) of the solution formulation to the tablet formulation; therefore the lowest dose available in the tablet formulation (250 mg) was selected.

DETAILED DESCRIPTION:
This is an open-label (volunteer and study staff will know the identity of the assigned treatment) study of two abiraterone acetate suspension formulations, compared to the abiraterone acetate tablet formulation in healthy volunteers. Approximately 30 healthy volunteers will participate in this study. Each volunteer will be randomly assigned to 1 of 6 possible treatment sequences. The study consists of a screening phase (within 21 days before the first study drug administration of the first period); an open-label treatment phase consisting of 3 single dose treatment periods; and end-of-study or withdrawal assessments done upon completion of the 72-hour (Day 4 of Period 3, or upon withdrawal) sampling to evaluate how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time. A 7- to 14-day washout period will separate the study drug administrations. The duration of participation in the study for an individual healthy volunteer will be from 41 days to a maximum of 55 days (including screening). Safety will be monitored. Volunteers will receive a 250 mg dose of abiraterone acetate as a tablet, suspension Formulation 1, and suspension Formulation 2 according to their treatment sequence. Abiraterone acetate tablets must be swallowed whole and not chewed, divided, dissolved or crushed and will be taken with 240 mL of noncarbonated water. For the suspensions, the volunteer will drink the contents of the vial. The vial will be rinsed with 10 mL of water, and the volunteer will be asked to drink the rinse water.

ELIGIBILITY:
Inclusion Criteria:

* Having signed an informed consent document
* Agreeing to use an adequate contraception method, as deemed appropriate by the investigator (e.g., vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Body mass index (weight [kg]/height2 [m]2) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Blood pressure (after the volunteer is sitting for 5 minutes) between 90 and 140 mm Hg systolic, inclusive, and no higher than 90 mm Hg diastolic during screening Days -21 to Day -1
* Having a 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function
* Morphology consistent with healthy cardiac conduction and function

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the volunteer or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or at admission to the study center as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs or 12-lead ECG at screening or at admission to the study center as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, within 14 days before the first dose of the study drug is scheduled
* History of, or a reason to believe a volunteer has a history of drug or alcohol abuse within the past 2 years

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Levels of study drug | Up to 55 days

SECONDARY OUTCOMES:
Vital signs evaluations | Up to 55 days
Adverse events | Up to 55 days
Clinical laboratory findings, based on blood and urine tests | Up to 55 days
Physical examination evaluations | Up to 55 days
Electrocardiogram changes | Up to 55 days

CONTACTS AND LOCATIONS:
Overall Officials: Cougar Biotechnology, Inc. Clinical Trial, Study Director — Cougar Biotechnology, Inc.